CLINICAL TRIAL: NCT02294370
Title: Glucose Excursions at Early Stages of Diabetes, MOSAIC Prospective Study
Brief Title: Variation of Glucose Values at Early Stages of Diabetes - Continuous Glucose Monitoring
Status: Completed | Type: Observational
Sponsor: Folkhälsan Researech Center (Other)
Collaborators: Medtronic (Industry); University of Padova (Other); Universidad Politecnica de Madrid (Other); University of Pavia (Other); Fondazione Salvatore Maugeri (Other); Asociación Española Para el Desarrollo de la Epidemiologia Clínica (Unknown); Lund University (Other); Soluciones Tecnologias para la Salud y el Bienestar SA (Unknown); National Technical University of Athens (Other)
Responsible Party: Sponsor
Other Study IDs: Botnia012014
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: type 2 diabetes; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- subjects at the early stages of diabetes: Subjects at the early stages of diabetes, individuals with impaired glucose tolerance (IGT, 2h plasma glucose during oral glucose tolerance test >7.8-11.1 mmol/l (n=50) or with type 2 diabetes (fasting plasma glucose > 7.0 mmol/l and/or 2h plasma glucose > 11.1 mmol/l on two occasions, or both criteria fulfilled in same oral glucose tolerance test while not pregnant, n=50) with short duration (<3 years)

SUMMARY:
This study aims at improving the prediction of type 2 diabetes among high-risk individuals by examining glucose excursion patterns in subjects with impaired glucose tolerance. In addition, this study will show whether the currently used diagnostic test could be replaced by an easier and less expensive method.

DETAILED DESCRIPTION:
Type 2 diabetes is a chronic disease of glucose metabolism leading to various disabling conditions. The onset of type 2 diabetes is a gradual shift from normal to abnormal, giving rarely noticeable symptoms at its early stages or even in later stages when damage has already been caused. Due to the gradual onset, the diagnosis is often delayed, and as much as half of the asymptomatic patients remain undetected. The diagnostic criteria for diabetes are based on artificial boundaries reflecting the risk of complications related to diabetes. The golden standard of diagnosis of diabetes is a 2 hours oral glucose tolerance test, which is both time consuming and costly. This study aims at improving the prediction of type 2 diabetes among high-risk individuals by examining glucose excursion patterns in subjects with impaired glucose tolerance. In addition, this study will show whether the currently used diagnostic test could be replaced by an easier and less expensive method.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with impaired glucose tolerance (2h plasma glucose during oral glucose tolerance test >7.8-11.1 mmol/l, n=50) or with type 2 diabetes (fasting plasma glucose > 7.0 mmol/l and/or 2h plasma glucose > 11.1 mmol/l on two occasions, or both criteria fulfilled in the same oral glucose tolerance test while not pregnant, n=50) with short duration (<3 years); 40 from Padova University Hospital, 60 from the Botnia Study or the PPP (Prevalence, Prediction, Prevention)-Botnia Study in Finland.
* Age 40-75 years

Exclusion Criteria:

* Medication with: insulin, glucagon-like peptide-1 (GLP-1)-analogues, sulphonylureas, oral corticosteroids, thyreostatic agents or thyroid hormone, luteinizing-hormone-releasing hormone (LHRH) analogues
* Pregnancy
* Known changes in retinal fundus photographs
* Known, microalbuminuria
* HbA1c >8%
* Fasting plasma glucose >10 mmol/l
* Medication with metformin, glitazones, gliptins (or acarbose) is allowed but gliptins and acarbose need to be stopped 2 days before testing and during the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with impaired glucose tolerance (2h plasma glucose during oral glucose tolerance test >7.8-11.1 mmol/l, n=50) or with type 2 diabetes (fasting plasma glucose > 7.0 mmol/l and/or 2h plasma glucose > 11.1 mmol/l on two occasions, or both criteria fulfilled in the same oral glucose tolerance test while not pregnant, n=50) with short duration (<3 years); 40 from Padova University Hospital, 60 from the Botnia Study or the PPP-Botnia Study in Finland. The Botnia Study and the PPP-Botnia Study are population based studies investigating type 2 diabetes in western Finland.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2013-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
glucose levels in tissue fluid | continuous monitoring for 1 week
  continuous glucose monitoring system

SECONDARY OUTCOMES:
capillary glucose | 4 times a day for 1 week
  for the calibration of the continuous glucose monitoring system

CONTACTS AND LOCATIONS:
Overall Officials: Tiinamaija Tuomi, MD,lecturer, Principal Investigator — Folkhalsan
Locations (1):
- Folkhälsan Research Center, Helsinki, Finland

REFERENCES:
- [Background] Soliman A, DeSanctis V, Yassin M, Elalaily R, Eldarsy NE. Continuous glucose monitoring system and new era of early diagnosis of diabetes in high risk groups. Indian J Endocrinol Metab. 2014 May;18(3):274-82. doi: 10.4103/2230-8210.131130. PMID 24944918
- [Background] Wang C, Lv L, Yang Y, Chen D, Liu G, Chen L, Song Y, He L, Li X, Tian H, Jia W, Ran X. Glucose fluctuations in subjects with normal glucose tolerance, impaired glucose regulation and newly diagnosed type 2 diabetes mellitus. Clin Endocrinol (Oxf). 2012 Jun;76(6):810-5. doi: 10.1111/j.1365-2265.2011.04205.x. PMID 21854404